CLINICAL TRIAL: NCT02584426
Title: Subcutaneous Injection and Ultrasonic Dispersion of Cefazolin Into Chronic Pelvic-Region Pressure Ulcers in Persons With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, William A. Bauman, M.D., Research Center Director, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAU-15-043
Record Dates: First submitted 2015-10-15; First posted 2015-10-22 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Spinal Cord Injury; Chronic Pressure Ulcers
Keywords: Cefazolin
MeSH Terms: conditions — Spinal Cord Injuries

ARMS (2):
- Cefazolin Treatment (Experimental): Subjects will receive antibiotic treatment with phonophoresis (i.e., hypodermoclysis) during test 1, and will be given standard of care for 8 weeks.
  Interventions: Device: Ultrasonic Distribution of Cefazolin
- Standard of Care Control (No Intervention): Subjects will not receive intervention and will receive standard of care for 8 weeks.

INTERVENTIONS:
Device: Ultrasonic Distribution of Cefazolin
  Arms: Cefazolin Treatment

SUMMARY:
Pressure ulcers (PU) are skin breakdowns that often form after blood flow in the skin is reduced from prolonged and repeated exposure to externally applied forces. As many as 85% of individuals with a spinal cord injury (SCI) report the occurrence of at least 1 PU since being injured. Despite the increasing attention and emphasis on prevention, PUs still represent a major health risk for persons with SCI. PUs and other skin breakdowns are at risk for becoming infected; it is not uncommon for many different types of "bugs" to be found in the wound. It has been assumed that the presence of these organisms did not impede wound healing or skin graft survival. The current proposal will use a new type of procedure that involves the direct injection of an antibiotic (in saline) into the skin beneath the wound; it is then distributed throughout the wound using a second device that uses sound waves. The study will determine if the antibiotic treatment and the standard of care improves the rate wound closure compared to the standard of care alone in persons with SCI and a chronic pelvic-region PU.

DETAILED DESCRIPTION:
Persons with spinal cord injury (SCI) are at increased risk of developing a Stage III or IV (full-thickness) pressure ulcer (PU). These wounds are associated with a tremendous personal and financial cost. An intervention that proves efficacious in the facilitation of healing this chronic medical condition would be of enormous medical, social, and economic benefit to persons with SCI and other cohorts with a difficult to heal PUs. From preliminary studies, it appears that hypodermoclysis (i.e., an interstitial infusion) with an antibiotic (i.e., cefazolin; a first generation cephalosporin) and subsequent dispersion with ultrasound throughout the wound recently has been shown in preliminary work to be efficacious in the treatment of infection, both recognized pathogenic organisms and those that have colonized the wound bed), which then appears to facilitate wound closure and success of standard surgical intervention. This approach to wound care represents a paradigm shift because previously it was assumed that nonpathogenic organism did not impede wound healing or skin graft survival. The investigators will test this novel approach to wound healing in persons with SCI who have a chronic PU of the pelvic region.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 to 79;
2. Chronic (e.g., duration of injury at least 6 months), stable SCI (regardless of level of neurological lesion);
3. American Spinal Injury Association Impairment Scale (AIS) designation of A or B with no sensation in the pelvic region;
4. At least one Stage III or IV PU in the pelvic region (e.g., ischial or trochanteric regions) that has not shown signs of healing for a period of at least 1 month;
5. At least one Stage III or IV PU in the pelvic region greater than 100 cm2 in surface area; and,
6. Hemoglobin A1C ≤7.0%.

Exclusion Criteria:

1. Persons who are candidates for or elect to have reconstructive flap surgery of the PU;
2. Unresolved osteomyelitis diagnosed by clinical impression and supported by one or more of the following: 1) history and examination of the pressure ulcer (i.e., visible bone), 2) bone contact on sterile probe, 3) bone that has lost its normal consistency, 4) magnetic resonance imaging, or 5) open bone biopsy;
3. Hemoglobin A1C >7.0%;
4. Psychopathology (documentation in the medical record or history of self-abusive behavior specific to PU healing which may or may not include major or minor psychiatric illness (that may conflict with the study objectives;
5. Acute illness or systemic infection;
6. Allergy to cefazolin;
7. Allergy to penicillin;
8. History of clinically significant or uncontrolled cardiac disease, including congestive heart failure, angina, myocardial infarction, arrhythmia, including New York Heart Association functional classification of 3;
9. Previously diagnosed active malignant disease;
10. Suspicion of skin cancer at the PU site (i.e., clinical evaluation is currently on-going);
11. Life expectancy less than 12 months;
12. Nephrosis, hemodialysis or chronic ambulatory peritoneal dialysis therapy;
13. Moderate to high dose glucocorticoid administrations (i.e., ≥ 40 mg prednisone or equivalent steroid dose) within the past 3 months;
14. Diminished mental capacity;
15. Inability or unwillingness of subject to provide informed consent; or,
16. Pregnancy or women who may become pregnant during the course of the study, or those who are nursing.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Percent Change in Surface area of a Chronic Pelvic Pressure Ulcer (PU) at 4 Weeks | 4 weeks
  1. To determine the percent change in surface area of a chronic pelvic region pressure ulcer (PU) 4 weeks after hypodermoclysis with antibiotic treatment and ultrasonic dispersion compared to standard of care.

SECONDARY OUTCOMES:
Percent Change in Surface area of a Chronic Pelvic Pressure Ulcer (PU) at 8 Weeks | 8 weeks
  2. To determine the percent change in surface area of a chronic pelvic region PU 8 weeks after hypodermoclysis with antibiotic treatment and ultrasonic dispersion compared to standard of care.

CONTACTS AND LOCATIONS:
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided